CLINICAL TRIAL: NCT02439619
Title: TechCare: Mobile-AssessmenT and ThErapy for PsyCHosis: An Intervention for Clients Within the EArly InteRvention SErvice
Acronym: TechCare
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lancashire Care NHS Foundation Trust (Network)
Collaborators: University of Central Lancashire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TechCare-LCFT
Record Dates: First submitted 2015-05-05; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Feasibility Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Feasibility Trial (Experimental)
  Interventions: Other: TechCare

INTERVENTIONS:
Other: TechCare — The TechCare software is being developed specifically for use on a touch screen mobile phone. The mobile application will alert participants through notifications and ask a number of questions. Based on participant responses the app will provide a CBT based response to individuals or the service users preferred multimedia such as music, images and videos.

SUMMARY:
The aim of the project is to conduct a feasibility study of the mobile phone application "TechCare" for individuals with psychosis in the North West of England.

DETAILED DESCRIPTION:
This feasibility study will follow the NIHR guidance on feasibility study design (NIHR, 2014) and will consist of both qualitative and quantitative components. The study will run across three strands as follows 1) Qualitative work & Systematic review 2) Test run and Intervention refinement 3) Feasibility trial.

ELIGIBILITY:
Inclusion Criteria:

* Each client must be accepted into the Psychosis Group of the Lancashire Early Intervention Service.
* Ages 18 - 35 years
* Medication stable for previous two months
* Clients must be currently stable-The Lancashire Early Intervention Team uses a traffic light system to indicate current symptomatology and risks of each client. For this study we will use only clients with a Green Light, signifying that they are currently stable.
* A score of 3 or more on positive symptoms on the PANSS
* Minimum score of 1 on the Calgary depression scale.

Exclusion Criteria:

* Drug induced psychosis
* An acquired brain injury or learning disability
* Clients who are undergoing assessment, not formally diagnosed and accepted into the service.
* Lacking capacity for informed consent.
* Ultra High Risk of Developing Psychosis Group (i.e. Prodromal, not first episode)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability | 36 months
  We will measure feasibility and acceptability by exploring whether appropriate individuals can be identified and recruited to an open trial of TechCare; whether TechCare is an acceptable intervention for individuals with psychosis and what measures will be important for assessing the impact of TechCare on delusions and low mood in psychosis.

SECONDARY OUTCOMES:
Psychopathology on The Positive and Negative Syndrome Scale (PANSS) | 24 months
  The 30- item PANSS, is a clinician administered 30 item semi structured interview which provides balanced representation of positive symptoms and negative symptoms and gauges their relationship to one another and to global/general psychopathology
Psychopathology on The Psychotic Symptom Rating Scales (PSYRATS) | 24 months
  The PSYRATS is a semi-structured interview measuring dimensions of delusions and hallucinations.
Satisfaction with CBT therapy on the CHoice of Outcome In Cbt for psychosEs | 24 months
  This is an outcome measure which reflects the aims of cognitive behavioural therapy for psychosis and the priorities of service users.
Mental wellbeing on the Warwick-Edinburgh Mental Well Being Scale (WEMWBS) | 24 months
  The WEMWBS is a measure of mental wellbeing which focuses entirely on positive aspects of mental health.
Measure of core beliefs regarding self and others on the Brief Core Schema Scale | 24 months
  This is a 24 item measure of core beliefs regarding self and others. It is a nine item scale which allows for the quantitative and subjective dimension of depression in schizophrenia.
Depression on the Calgary depression scale | 24 months
  The CDS was developed to measure the level of depression in schizophrenia. It is a nine item scale which allows for the quantitative and subjective dimension of depression in schizophrenia.
Work and social functioning on The Work and Social Adjustment Scale | 24 months
  This is a five item measure of perceived impairment in five areas: work, home management, social life, private leisure and relationships
Quality of life on the EuroQoL-5 Dimensions EQ5-D | 24 months
  the measure is standardised instrument looking at quality of life across five health domains (mobility, self-care, usual activities, pain/discomfort and anxiety/depression).

CONTACTS AND LOCATIONS:
Overall Officials: Imran B Chaudhry, MBBS MD, Principal Investigator — Lead Consultant Psychiatrist, Lancashire Care Early Intervention Service & Hon Clinical Professor Adult Psychiatry University of Manchester; Nusrat Husain, MBBS MD, Principal Investigator — Reader in Psychiatry University of Manchester, Director Research Global Health Manchester Academic Health Sciences Centre & Consultant Psychiatrist Lancashire Care Early Intervention Service; James Kelly, DClinPsych, Principal Investigator — Lancashire Care NHS Foundation Trust Early Intervention Service
Locations (1):
- Lancashire Care NHS Foundation Trust, Preston, Lancashire, United Kingdom

REFERENCES:
- [Derived] Gire N, Caton N, McKeown M, Mohmed N, Duxbury J, Kelly J, Riley M, J Taylor P, Taylor CDJ, Naeem F, Chaudhry IB, Husain N. 'Care co-ordinator in my pocket': a feasibility study of mobile assessment and therapy for psychosis (TechCare). BMJ Open. 2021 Nov 16;11(11):e046755. doi: 10.1136/bmjopen-2020-046755. PMID 34785541